CLINICAL TRIAL: NCT00451919
Title: Sickle-Cell Disease: Neuroimaging and Cognitive Decline
Brief Title: The Link Between Anemia and Deficits in Memory and Attention in Individuals With Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: University of California, San Francisco (Other)
Other Study IDs: 375; K01HL073152 (NIH)
Record Dates: First submitted 2007-03-23; First posted 2007-03-26 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2013-10

CONDITIONS: Sickle Cell Disease
Keywords: MRI; Neuropsychology
MeSH Terms: conditions — Anemia, Sickle Cell

SUMMARY:
Sickle cell disease is an inherited blood disorder that affects red blood cells (RBCs). People with sickle cell disease frequently experience anemia, or a low number of RBCs. RBCs are responsible for carrying oxygen to the brain and other body tissues that need oxygen to function properly. The purpose of this study is to determine what changes, which were possibly caused by anemia, exist in the brains of individuals with sickle cell disease.

DETAILED DESCRIPTION:
The role of RBCs is to carry oxygen from the lungs to the brain and other body tissues. Individuals with anemia have unusually low numbers of RBCs. They also often have difficulty concentrating and remembering information, which is likely caused by a reduced oxygen supply to the brain. Previous research has shown that correcting anemia in patients without sickle cell disease improved their memory and attention. The purpose of this study is to examine any abnormal changes in the brains of individuals with sickle cell disease and to determine whether these changes are related to reduced memory and attention capabilities.

Participants will attend one study visit. During this visit, a brain magnetic resonance image (MRI) will be performed while participants complete neuropsychological tests that measure memory, attention, and organizational ability. There will be no follow-up visits.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sickle cell disease

Exclusion Criteria:

* Pregnancy
* Claustrophobia
* Mass lesion (e.g., meningioma, cyst, or spinal block)
* Need for life support constant monitoring
* Any unstable condition that is likely to require resuscitation
* Presence of a pacemaker or other iron-containing magnetic substances in the body

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall R. Rule, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States